CLINICAL TRIAL: NCT03880552
Title: Perineal Body Length and Perineal Lacerations During Delivery in Primigravid Patients
Brief Title: Perineal Body Length and Perineal Lacerations
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Pınar Kadirogulları, pınar kadiroğulları M.D, Department of Obstetrics and Gynecology, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: 2018.12.68
Record Dates: First submitted 2019-03-14; First posted 2019-03-19 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Perineal Laceration Involving Skin; Delivery; Trauma
Keywords: perineal laceration; obstetric trauma
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Primigravid women with singleton pregnancy at 35th week over — Primigravid women with singleton pregnancy at 35th week over; only observational study will be done in this group and the data will be recorded.

SUMMARY:
The aim of this study was to evaluate the relationship between perineal body length and perineal laceration risk in primigravid patients.

Primigravid women with singleton pregnancies in the first stage of labor at the 35th week of gestation were included in the study. The peineal body length of the patients was measured by the same physician.

DETAILED DESCRIPTION:
After 35 weeks of gestation, nulliparous women with single gestation were included in the study and genital hiatus and perineal body measurements were taken.

The presence and degree of perineal laceration after birth were determined. Correlation of genital hiatus and perineal body measurements with perineal laceration risk were evaluated.

After birth, vaginal laceration, oxytocin use, fetal birth weight, the presence of episiotomy were recorded.

ELIGIBILITY:
Inclusion Criteria:

-Primigravid women with singleton pregnancy at over 35th week

Exclusion Criteria:

* the story of operative vaginal birth;
* caesarean section;
* breech presentation;
* those with a history of anorectal surgery or trauma

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Meet the criteria of inclusion in our hospital for birth,The study was planned for women with singleton pregnancies of 35 weeks or more.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Perineal body length | during delivery
  The length of the perineal body will be measured in centimeters.
perineal laceration | during delivery
  Laceration measurement 1.-2.-3.-4. degree. The measurement of laceration will be graded.
  1. st degree laceration is the tears formed in the vaginal epithelium and perineum skin.
  2. nd degree laceration includes perineal muscles. 3. Degree lacerations extend to the anal sphinkter complex. In the 4th degree laceration, the anal epithelium / rectal mucosa was also torn.

SECONDARY OUTCOMES:
genital hiatus length | during delivery
  The length of the genital hiatus will be measured in centimeters.

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni Sultan Süleyman Training and Research Hospital, Istanbul, Turkey (Türkiye)